CLINICAL TRIAL: NCT01883362
Title: A Phase II, Randomized Trial of Standard of Care, With or Without Midostaruin to Prevent Relapse Following Allogeneic Hematopoietic Stem Cell Transplantation in Patients With FLT3-ITD Mutated Acute Myeloid Leukemia
Brief Title: Standard of Care +/- Midostaurin to Prevent Relapse Post Stem Cell Transplant in Patients With FLT3-ITD Mutated AML
Acronym: RADIUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPKC412AUS23
Record Dates: First submitted 2013-03-25; First posted 2013-06-21 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; AML; FLT3-ITD; midostaurin; PKC412; allogeneic hematopoeitic stem cell tranplant; SCT; HSCT; CR1; adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care with Midostaurin (Experimental): Patients received standard of care in the post stem cell transplant (SCT) setting in addition to Midostaurin 50mg twice a day for 12 months (cycles).
  Interventions: Drug: Midostaurin
- Standard of Care (Active Comparator): Patients received standard of care alone in the post SCT setting
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Midostaurin — Midostaurin was supplied in 25mg soft gelatin capsule taken orally twice a day for 28 days of each cycle. Patients will be treated for 12 cycles.
  Other Names: PKC412
  Arms: Standard of Care with Midostaurin
Other: Standard of Care — Standard of Care was not defined per protocol. The investigator prescribed based on the commonly used medications given in the post SCT setting.
  Arms: Standard of Care

SUMMARY:
To determine if the addition of midostaurin (PKC412) to Standard of Care (SOC) therapy reduces relapse in FLT3-ITD mutated AML patients receiving an allogenetic hematopoietic stem cell transplant,

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age
* Patients with ECOG Performance Status of ≤ 2
* Patients with a documented unequivocal diagnosis of AML according to WHO 2008 classification (>20% blasts in the bone marrow), excluding M3 (acute promyelocytic leukemia).
* Patients with a documented FLT3 ITD mutation, determined by local laboratory for eligibility (historical tissue will be requested for central analysis confirmation)
* Patients who undersent allogeneic HSCT in CR1 from a matched related or matched unrelated donor. All of the following criteria had to be met: HLA typing to include available 8/8 or 7/8 allele HLA matched donor (at A,B,C, DRB1) Single allelic mismatch allowed
* Patients who had received a conditioning regimen which included one of the following:

Busulfan/Fludarabine (Bu/Flu) Busulfan (16 mg/kg PO or 12.8 mg/kg IV) Fludarabine (120-180 mg/m2) Fludarabine / Melphalan (Flu/Mel) Fludarabine (120-180 mg/m2) Melphalan (≤ 150 mg/m2) Busulfan/Cyclophosphamide (Bu/Cy) Busulfan (16 mg/kg PO or 12.8 mg/kg IV) Cyclophosphamide (120 mg/kg) Cyclophosphamide/Total Body Irradiation (Cy/TBI) Cyclophosphamide (120 mg/kg) TBI (1200-1420 cGy)

• Recovery of counts by day 42 and was able to start midostaurin by day 60 post-HSCT (first dose of midostaurin to start no earlier than 28 days post-HSCT); ANC >1000µL, platelets ≥20,000 without platelet transfusion

Exclusion Criteria:

Patients eligible for this study must not have met any of the following criteria:

* Patients who failed prior attempts at allogeneic HSCT
* Patients who had received an autologous transplant
* Patients with Acute GVHD Grade III-IV
* Patients with a known confirmed diagnosis of HIV infection or active viral hepatitis.
* Impaired cardiac function including any of the following:

  * Screening ECG with a QTc > 450 msec. If QTc > 450 and electrolytes were not within normal ranges, electrolytes should be corrected and then the patient rescreened for QTc.
  * Patients with congenital long QT syndrome
  * History or presence of sustained ventricular tachycardia
  * Any history of ventricular fibrillation or torsades de pointes
  * Bradycardia defined as HR. < 50 bpm
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Patients with myocardial infarction or unstable angina < 6 months prior to starting study
  * Congestive Heart Failure NY Heart Association class III or IV
  * Patients with an ejection fraction < 45% assessed by MUGA or ---ECHO within 28 days prior to starting study cycle 1 (of midostaurin or control group)
* Patients with any pulmonary infiltrate including those suspected to be of infectious origin (unless resolves to ≤ Grade 1 within screening timeframe)
* Patient required treatment with strong CYP3A4 inhibitors or moderate or strong CYP3A4 inducers other than those required for GVH or infection prophylaxis or treatment

Pregnant or nursing (lactating) women, or women of child-bearing potential, must have used highly effective methods of contraception during dosing and for 30 days after treatment completion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Elliott, MD, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (18):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - University of California at Los Angeles Oncology, Los Angeles, California
  - SCRI- Colorado Blood Cancer Institute, Denver, Colorado
  - H Lee Moffitt Cancer Center and Research Institute Oncology, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Karmanos Cancer Institute Karmanos - Wayne State, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School Of Medicine-Siteman Cancer Ctr Washington U School of Med, St Louis, Missouri
  - Hackensack University Medical Center Hackensack Univ Med Ctr (32), Hackensack, New Jersey
  - University of North Carolina at Chapel Hill University of North Carolina 6, Chapel Hill, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Tennessee Oncology Sarah Cannon Research Inst., Nashville, Tennessee
  - Vanderbilt Univeristy Oncology, Nashville, Tennessee
  - Baylor Health Care System/Sammons Cancer Center Oncology, Dallas, Texas
  - Texas Transplant Physicians Group Oncology 2, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center Oncology, Seattle, Washington
- Novartis Investigative Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Maziarz RT, Levis M, Patnaik MM, Scott BL, Mohan SR, Deol A, Rowley SD, Kim DDH, Hernandez D, Rajkhowa T, Haines K, Bonifacio G, Rine P, Purkayastha D, Fernandez HF. Midostaurin after allogeneic stem cell transplant in patients with FLT3-internal tandem duplication-positive acute myeloid leukemia. Bone Marrow Transplant. 2021 May;56(5):1180-1189. doi: 10.1038/s41409-020-01153-1. Epub 2020 Dec 7. PMID 33288862

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Started | 30 | 30
Completed | 14 | 16
Not Completed | 16 | 14
Not completed — Adverse Event | 1 | 8
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Administrative problems | 4 | 1
Not completed — Relapse | 4 | 2
Not completed — Randomized, not treated | 1 | 1
Period: Post Treatment Follow-up
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Started | 26 | 27
Completed | 10 | 13
Not Completed | 16 | 14
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 4
Not completed — Administrative problems | 2 | 0
Not completed — Death | 8 | 4
Not completed — Relapse | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care With Midostaurin | Standard of Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (13.68) | 46.0 (11.08) | 48.4 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 16 | 18 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 27 | 27 | 54
  Black | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Other | 1 | 2 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.9934 (7.11368) | 26.6400 (5.27475) | 26.8101 (6.17055)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Relapse Free Survival (RFS) up to 18 Months Post Transplant (Full Analysis Set) by Kaplan-Meier Analysis
Description: Relapse-free survival assesses the clinical benefit of remaining in remission free from relapse or death due to the disease. It was defined as the time from transplant to relapse or death due to the disease. Relapse following complete response was defined as reappearance of leukemic blasts in the peripheral blood or finding more than 5% blasts in the bone marrow.
Time Frame: date of transplant up to 18 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 30 | 30
proportion of participants
  6 months | 0.93 [0.75 to 0.98] | 0.93 [0.74 to 0.98]
  12 months | 0.80 [0.59 to 0.91] | 0.93 [0.74 to 0.98]
  18 months | 0.76 [0.54 to 0.88] | 0.89 [0.69 to 0.96]
Statistical Analysis 1: Comparison: Standard of Care With Midostaurin vs Standard of Care; Test type: Superiority; p = 0.2655, Log Rank; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.12 to 1.86]

2. Secondary Outcome: Proportion of Participants With Relapse Free Survival (RFS) - Time From Randomization up to 18 Months (Full Analysis Set) by Kaplan-Meier Analysis
Description: as for outcome 1
Time Frame: Randomization to 18 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 30 | 30
Proportion of participants
  6 months | 0.93 [0.75 to 0.98] | 0.93 [0.74 to 0.98]
  12 months | 0.80 [0.59 to 0.91] | 0.93 [0.74 to 0.98]
  18 months | 0.76 [0.54 to 0.88] | 0.85 [0.64 to 0.94]
Statistical Analysis 1: Comparison: Standard of Care With Midostaurin vs Standard of Care; Test type: Superiority; p = 0.4297, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.17 to 2.14]

3. Secondary Outcome: Proportion of Participants With Relapse Free Survival (RFS) - Time From Randomization up to 24 Months(Full Analysis Set) by Kaplan-Meier Analysis
Description: DFS was defined as the time from transplant to relapse or death due to any cause. If a patient had more than 1 event (e.g., relapse then death) then the earliest date was taken into account.
Time Frame: date of transplant up to 24 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 30 | 30
Proportion of participants
  6 months | 0.90 [0.71 to 0.96] | 0.93 [0.74 to 0.98]
  12 months | 0.77 [0.56 to 0.89] | 0.89 [0.70 to 0.96]
  18 months | 0.69 [0.48 to 0.83] | 0.85 [0.65 to 0.94]
  24 months | 0.69 [0.48 to 0.83] | 0.81 [0.61 to 0.92]
Statistical Analysis 1: Comparison: Standard of Care With Midostaurin vs Standard of Care; Test type: Superiority; p = 0.2424, Log Rank; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.20 to 1.52]

4. Secondary Outcome: Proportion of Participants With Relapse Free Survival (RFS) - Time From Transplant (Full Analysis Set) by Kaplan-Meier Analysis
Description: Relapse-free survival was defined as the time from transplant to relapse or death due to the disease 24 months post-transplant. If a patient had more than one event (e.g., relapse then death) then the earliest date was taken into account.
Time Frame: date of transplant up to 24 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 30 | 30
Proportion of participants
  6 months | 0.93 [0.75 to 0.98] | 0.93 [0.74 to 0.98]
  12 months | 0.80 [0.59 to 0.91] | 0.93 [0.74 to 0.98]
  18 months | 0.76 [0.54 to 0.88] | 0.89 [0.69 to 0.96]
  24 months | 0.76 [0.54 to 0.88] | 0.85 [0.64 to 0.94]
Statistical Analysis 1: Comparison: Standard of Care With Midostaurin vs Standard of Care; Test type: Superiority; p = 0.4297, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.17 to 2.14]

5. Secondary Outcome: Probability of Overall Survival - Date of Transplant up to 24 Months (Full Analysis Set) by Kaplan-Meier Analysis
Description: Overall survival was defined as the time from transplant to death due to any cause.
Time Frame: date of transplant up to 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 30 | 30
proportion of participants
  6 months | 0.96 [0.71 to 0.96] | 1.00 [1.00 to 1.00]
  12 months | 0.89 [0.56 to 0.89] | 0.89 [0.69 to 0.96]
  18 months | 0.76 [0.54 to 0.89] | 0.85 [0.65 to 0.94]
  24 months | 0.76 [0.54 to 0.89] | 0.85 [0.65 to 0.94]
Statistical Analysis 1: Comparison: Standard of Care With Midostaurin vs Standard of Care; Test type: Superiority; p = 0.3418, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.19 to 1.79]

6. Secondary Outcome: Probability of Non-relapse Mortality (NRM) - Date of Transplant up to 24 Months (Full Analysis Set) by Kaplan-Meier Analysis
Description: Non-relapse mortality (NRM) was defined as the time from transplant to death due to reasons other than relapse/progressive disease
Time Frame: date of transplant up to 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 30 | 30
proportion of participants
  6 months | 0.96 [0.77 to 0.99] | 1.00 [1.00 to 1.00]
  12 months | 0.96 [0.77 to 0.99] | 0.96 [0.76 to 0.99]
  18 months | 0.92 [0.71 to 0.98] | 0.96 [0.76 to 0.99]
  24 months | 0.92 [0.71 to 0.98] | 0.96 [0.76 to 0.99]
Statistical Analysis 1: Comparison: Standard of Care With Midostaurin vs Standard of Care; Test type: Superiority; p = 0.4169, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.09 to 2.74]

7. Secondary Outcome: FLT3-ITD Mutation Status Centrally in Archived Material From Diagnosis (if Available) Including Mutant:Wild Type Ratio.
Description: Unable to retrieve a sufficient amount of archived samples to perform an analysis therefore the study was not able to verify the FLT3-ITD mutation status
Time Frame: up to 24 months from date of transplannt or at study completion
Population: Insufficient amount of samples to perform analysis
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Plasma Pharmacokinetics (PK) of Midostaurin and the Metabolites: CGP62221 and CGP52421: Pre-dose Levels
Description: Pre-dose levels (Cmin) will be directly determined from raw plasma concentration-time data. Values below the lower limit of quantification (LLOQ) will be treated as zero in any calculations of summary statistics.
Time Frame: Pre-dose on days 1 and 15 of Cycle 1, on day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: number of samples available differed across time points
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- PKC412: Patients received standard of care in the post stem cell transplant (SCT) setting in addition to Midostaurin 50mg twice a day for 12 months (cycles).
- Metabolite CGP52421: Metabolite of PKC412 (CGP52421)
- Metabolite CGP62221: Metabolite of PKC412 (CGP62221)
Arm/Group | PKC412 | Metabolite CGP52421 | Metabolite CGP62221
Number analyzed (Participants) | 29 | 29 | 29
ng/ml
  Visit 2,Cycle1,Day 1: number analyzed (Participants) | 27 | 27 | 27
  Visit 2,Cycle1,Day 1 | 17.46 (76.806) | 0.00 (0.000) | 16.89 (61.212)
  Visit 4,Cycle1, Day 15: number analyzed (Participants) | 28 | 28 | 29
  Visit 4,Cycle1, Day 15 | 932.46 (770.597) | 1572.69 (684.955) | 906.57 (747.836)
  Visit 5,Cycle2,Day 1: number analyzed (Participants) | 26 | 26 | 26
  Visit 5,Cycle2,Day 1 | 769.92 (485.353) | 1768.77 (849.580) | 779.90 (400.244)
  Visit 6,Cycle3,Day 1: number analyzed (Participants) | 20 | 20 | 20
  Visit 6,Cycle3,Day 1 | 907.20 (528.017) | 2051.55 (765.758) | 929.45 (311.841)
  Visit 7,Cycle4,Day 1: number analyzed (Participants) | 20 | 20 | 20
  Visit 7,Cycle4,Day 1 | 548.45 (459.294) | 1707.15 (810.143) | 714.00 (610.925)
  Visit 8,Cycle5,Day 1: number analyzed (Participants) | 20 | 20 | 20
  Visit 8,Cycle5,Day 1 | 525.73 (255.032) | 1742.85 (658.905) | 722.00 (320.977)
  Visit 9,Cycle6,Day 1: number analyzed (Participants) | 21 | 21 | 21
  Visit 9,Cycle6,Day 1 | 519.10 (328.032) | 1757.86 (685.740) | 763.86 (408.290)
  Visit 10,Cycle 7 Day 1: number analyzed (Participants) | 20 | 20 | 20
  Visit 10,Cycle 7 Day 1 | 754.95 (497.976) | 1717.35 (720.259) | 780.65 (424.200)
  Visit 11,Cycle 8 Day 1: number analyzed (Participants) | 19 | 19 | 19
  Visit 11,Cycle 8 Day 1 | 537.95 (229.529) | 1787.21 (733.162) | 774.84 (326.583)
  Visit 12,Cycle 9 Day 1: number analyzed (Participants) | 17 | 17 | 17
  Visit 12,Cycle 9 Day 1 | 571.76 (311.764) | 1889.76 (678.435) | 850.47 (328.411)
  Visit 13,Cycle 10 Day 1: number analyzed (Participants) | 18 | 18 | 18
  Visit 13,Cycle 10 Day 1 | 643.07 (452.268) | 1836.50 (632.894) | 851.38 (347.311)
  Visit 14,Cycle 11 Day 1: number analyzed (Participants) | 18 | 18 | 18
  Visit 14,Cycle 11 Day 1 | 718.22 (538.208) | 1857.33 (868.406) | 983.94 (801.361)
  Visit 15,Cycle 12 Day 1: number analyzed (Participants) | 17 | 17 | 17
  Visit 15,Cycle 12 Day 1 | 564.69 (410.156) | 1706.29 (643.326) | 763.60 (387.685)

9. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 12.5 months (treatment duration ranged from 0.2 to 11.5 months). Deaths post treatment survival follow up were collected after the on treatment period, up to approximately 51 months.
Time Frame: approx. 12.5 months, approx. 51 months
Population: Clinical Database Population: all treated patients
Measure: Number; unit: Participants
Arm/Group | Standard of Care With Midostaurin | Standard of Care
Number analyzed (Participants) | 30 | 30
Participants
  Total Deaths | 8 | 4
  Deaths on-treatment | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 12.5 months (treatment duration ranged from 0.2 to 11.5 months).
Description: AE: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- ALL Patients: ALL Patients combined
Arm/Group | Standard of Care With Midostaurin | Standard of Care | ALL Patients
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30 | 1/60
Serious Adverse Events (participants affected / at risk) | 9/30 | 15/30 | 24/60
Other Adverse Events (participants affected / at risk) | 28/30 | 26/30 | 54/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care With Midostaurin (N=30) | Standard of Care (N=30) | ALL Patients (N=60)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 1
Myocarditis (Cardiac disorders) | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 4
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Chills (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 2 | 4
Chronic graft versus host disease in intestine (Immune system disorders) | 1 | 0 | 1
Chronic graft versus host disease in liver (Immune system disorders) | 1 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 1 | 2
Encephalitis (Infections and infestations) | 1 | 0 | 1
Enterovirus infection (Infections and infestations) | 0 | 1 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 1
Mycobacterium fortuitum infection (Infections and infestations) | 0 | 1 | 1
Nocardiosis (Infections and infestations) | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 2
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Amylase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Psychogenic seizure (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care With Midostaurin (N=30) | Standard of Care (N=30) | ALL Patients (N=60)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 10
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 5
Sinus tachycardia (Cardiac disorders) | 3 | 1 | 4
Tachycardia (Cardiac disorders) | 1 | 3 | 4
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 3
Cushingoid (Endocrine disorders) | 2 | 1 | 3
Hypothyroidism (Endocrine disorders) | 2 | 1 | 3
Dry eye (Eye disorders) | 5 | 5 | 10
Lacrimation increased (Eye disorders) | 1 | 2 | 3
Vision blurred (Eye disorders) | 4 | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 7
Constipation (Gastrointestinal disorders) | 4 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 9 | 4 | 13
Dry mouth (Gastrointestinal disorders) | 5 | 4 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 4
Flatulence (Gastrointestinal disorders) | 3 | 0 | 3
Nausea (Gastrointestinal disorders) | 19 | 5 | 24
Oral pain (Gastrointestinal disorders) | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 3
Vomiting (Gastrointestinal disorders) | 20 | 5 | 25
Asthenia (General disorders) | 1 | 2 | 3
Catheter site pain (General disorders) | 2 | 0 | 2
Chest discomfort (General disorders) | 0 | 2 | 2
Chest pain (General disorders) | 2 | 0 | 2
Chills (General disorders) | 1 | 3 | 4
Fatigue (General disorders) | 7 | 7 | 14
Malaise (General disorders) | 0 | 2 | 2
Mucosal inflammation (General disorders) | 0 | 2 | 2
Oedema peripheral (General disorders) | 6 | 10 | 16
Pain (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 3 | 4 | 7
Graft versus host disease (Immune system disorders) | 2 | 1 | 3
Graft versus host disease in eye (Immune system disorders) | 0 | 2 | 2
Graft versus host disease in skin (Immune system disorders) | 2 | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 4 | 4
Folliculitis (Infections and infestations) | 0 | 2 | 2
Influenza (Infections and infestations) | 2 | 0 | 2
Rhinovirus infection (Infections and infestations) | 2 | 1 | 3
Sinusitis (Infections and infestations) | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 9
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 5 | 6 | 11
Aspartate aminotransferase increased (Investigations) | 5 | 7 | 12
Blood alkaline phosphatase increased (Investigations) | 3 | 5 | 8
Blood bilirubin increased (Investigations) | 2 | 1 | 3
Blood cholesterol increased (Investigations) | 0 | 2 | 2
Blood creatinine increased (Investigations) | 3 | 3 | 6
Blood triglycerides increased (Investigations) | 0 | 2 | 2
Lipase increased (Investigations) | 1 | 2 | 3
Lymphocyte count decreased (Investigations) | 1 | 2 | 3
Neutrophil count decreased (Investigations) | 7 | 3 | 10
Platelet count decreased (Investigations) | 4 | 3 | 7
Transaminases increased (Investigations) | 0 | 2 | 2
Weight decreased (Investigations) | 2 | 3 | 5
White blood cell count decreased (Investigations) | 6 | 2 | 8
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Dizziness (Nervous system disorders) | 3 | 6 | 9
Dizziness postural (Nervous system disorders) | 2 | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 3 | 4
Headache (Nervous system disorders) | 8 | 5 | 13
Hyperaesthesia (Nervous system disorders) | 2 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 3
Tremor (Nervous system disorders) | 5 | 3 | 8
Anxiety (Psychiatric disorders) | 3 | 2 | 5
Depression (Psychiatric disorders) | 2 | 2 | 4
Insomnia (Psychiatric disorders) | 4 | 6 | 10
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 2 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 2
Renal failure (Renal and urinary disorders) | 1 | 2 | 3
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Melanocytic naevus (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 10
Rash (Skin and subcutaneous tissue disorders) | 5 | 6 | 11
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Hypertension (Vascular disorders) | 2 | 6 | 8
Hypotension (Vascular disorders) | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-07-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT01883362/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT01883362/SAP_001.pdf